CLINICAL TRIAL: NCT05054140
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate Efficacy, Safety, and Tolerability of IMU-838 in Patients With Progressive Multiple Sclerosis
Brief Title: Study to Evaluate Efficacy, Safety, and Tolerability of IMU-838 in Patients With Progressive Multiple Sclerosis
Acronym: CALLIPER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunic AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P2-IMU-838-PMS
Record Dates: First submitted 2021-09-02; First posted 2021-09-23 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis
Keywords: Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMU-838 (Experimental): IMU-838 as tablet; Administration: Oral - daily
  Interventions: Drug: IMU-838
- Placebo (Placebo Comparator): Matching placebo as tablet; Administration: Oral - daily
  Interventions: Drug: Placebo matching IMU-838

INTERVENTIONS:
Drug: IMU-838 — IMU-838 tablets
  Other Names: Vidofludimus calcium
  Arms: IMU-838
Drug: Placebo matching IMU-838 — Placebo matching IMU-838 tablets
  Other Names: Placebo Arm
  Arms: Placebo

SUMMARY:
Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate Efficacy, Safety, and Tolerability of IMU-838 in Patients with Progressive Multiple Sclerosis - CALLIPER

DETAILED DESCRIPTION:
This study will be a multicenter, randomized, double-blind, placebo-controlled study with a blinded Main Treatment Period (MT) and an Open Label Period (OLE) to evaluate the efficacy, safety, and tolerability of IMU838 in adult patients with PMS. The study will consist of the following periods:

Screening Period: Approximately 28 days Main Treatment Period: Up to 120 weeks (approximately 2 years) Open Label Extension Period: Up to approximately 8 years

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age 18 to 65 years (inclusive).
* EDSS score at screening between 3.0 to 6.5 (both inclusive)
* No evidence of relapse in the last 24 months before randomization, AND Patients diagnosed according to 2017 revised McDonald Criteria 1 and the 2013 revised classification of disease courses 2 as either

  1. SPMS inpatients showing evidence of Gd+MRI lesions (active SPMS) or without Gd+MRI lesions (non-active SPMS) in the last 12 months, OR
  2. PPMS
* Willingness and ability to comply with the protocol.
* Written informed consent given by the patient before the beginning of any study-related procedure.
* Documented evidence of disability progression not temporarily related to a relapse in the last 24 months before randomization, adjudicated by a central independent reviewer

Exclusion Criteria:

* Any disease other than MS that may better explain the signs and symptoms, including a history of complete transverse myelitis.
* Clinical signs or presence of laboratory findings suggestive for neuromyelitis optica (NMO) spectrum disorders or myelin oligodendrocyte glycoprotein (MOG)-associated encephalomyelitis (i.e.,presence of anti-NMO [aquaporin-4] antibodies or anti-MOG antibodies).
* Previous or current use of MS treatments lifelong, or within a pre-specified time period.
* Use of any investigational product within 8 weeks or 5 the respective PK half- life before the date of informed consent, whichever is longer, and throughout the study.For some investigational products, prolonged biological effects beyond 8 weeks should be considered.
* Positive test for severe acute respiratory syndrome coronavirus 2 (SARS- CoV-2) within14 days before randomization. In case of known SARS-CoV-2 infection, patients should be randomized no earlier than 14 days after 2 consecutive negative tests confirming virus negative status.The screening period can be extended for these patients to accommodate the required virus negativity.
* Positive IFN-gamma release assay (IGRA) for Mycobacterium tuberculosis at SV1.
* Positive hepatitis B virus (HBV) surface antigen, hepatitis B core antibody, positive hepatitis C virus (HCV) antibody, and/or HIV-antigen-antibody test at SV1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-01-07 (Estimated); Study Completion 2025-01-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of IMU-838 versus placebo | 120 weeks
  Annualized rate of percent brain volume change (PBVC) during MT period

SECONDARY OUTCOMES:
Efficacy of IMU-838 versus placebo | 120 weeks
  Annualized rate of change in brain parenchymal fraction (BPF) during MT Period
Efficacy of IMU-838 versus placebo in terms of disability worsening | 120 weeks
  Time to 24-week confirmed disability worsening based on expanded disability status scale (EDSS) during MT Period

OTHER OUTCOMES:
Safety IMU-838 versus placebo | 120 weeks
  Adverse events (AEs) and serious AEs (SAEs) during MT Period

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Fox, MD, Principal Investigator — Mellen Center for MS, Neurological Institute, Cleveland Clinic, Ohio
Locations (73):
- United States (8):
  - Dr. Sonia Kalirao, Coral Springs, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Prof. James Scott, Ormond Beach, Florida
  - Shepherd Center, Atlanta, Georgia
  - Consultants in Neurology, Ltd., Northbrook, Illinois
  - Dr. Daniel Becker, Lutherville, Maryland
  - Dr. Mirela Cerghet, Detroit, Michigan
  - University of New Mexico (UNM), MS Specialty Clinic, Albuquerque, New Mexico
- Bulgaria (19):
  - MHAT Pulse, Blagoevgrad
  - MHAT"Heart and Brain" EAD, Burgas
  - Dr. Maya Danovska, Pleven
  - Dr. Plamen Bozhinov, Pleven
  - UMHAT Pulmed, Plovdiv
  - Dr. Rositsa Krasteva, Rousse
  - Dr. Nikolay Georgiev, Shumen
  - MHAT Shumen, Shumen
  - Dr. Ivan Milanov, Sofia
  - MHAT Lyulin, Sofia
  - Dr. Rosen Ikonomov, Sofia
  - Dr. Penko Shotekov, Sofia
  - UMHAT Alexandrovska, Sofia
  - Dr. Kana Prinova, Sofia
  - Dr. Kosta Kostov, Sofia
  - MHAT Sveta Sofia, Sofia
  - UMHATSM N.I.Pirogov, Sofia
  - UMHAT Prof. Stoyan Kirkovich, Stara Zagora
  - Dr. Ara Kaprelyan, Varna
- Canada (2):
  - Montreal Neurological Inst., Montreal
  - The Ottawa Hospital Research Institute, Ottawa
- Fakultni nemocnice, Hradec Králové, Czechia
- Germany (4):
  - Datamed GmbH, Cologne
  - Klinik und Poliklinik für Neurologie, Universitätsklinikum Dresden, Dresden
  - Neuro Centrum Science GmbH, Erbach im Odenwald
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
- Moldova (3):
  - Dr. Stanislav Groppa, Chisinau
  - Dr. Mihail Gavriliuc, Chisinau
  - Dr. Olesea Odainic, Chisinau
- Netherlands (2):
  - Dr. Eva Strijibis, Amsterdam
  - Alrijne ziekenhuis, Leiderdorp
- North Macedonia (3):
  - Dr. Ana Doneva Skopje 1000, Skopje
  - Dr. Milcho Demerdziev, Skopje
  - Dr. Tatjana Boshkova, Skopje
- Poland (14):
  - Dr. Robert Bonek, Bydgoszcz
  - Dr. Maciej Maciejowski, Katowice
  - Dr. Janusz Zbrojkiewicz, Katowice
  - Dr. Elzbieta Jasinska, Kielce
  - Indywidualna Praktyka Lekarska Prof. Rejdak, Lublin
  - Dr. Marcin Nastaj, Lublin
  - Instytut Zdrowia, Oświęcim
  - Dr. Justyna Hryniewicz, Plewiska
  - Clinical Research Center, Poznan
  - EMC PL Certus, Poznan
  - NZOZ "Neuro-kard", Poznan
  - Dr. Marcin Ratajczak, Szczecin
  - Warszawska Klinika, Warsaw
  - EMC Instytut Medyczny, Wroclaw
- Romania (2):
  - Dr. Adriana Dulamea, Bucharest
  - Dr. Lacramioara Perju-Dumbrava, Cluj-Napoca
- Serbia (4):
  - Clinical Hospital Center Zemun, Belgrade
  - Military Medical Academy, Belgrade
  - Klinicki Centar Kragujevac, Kragujevac
  - Clinical center of Vojvodina, Novi Sad
- Ukraine (11):
  - Chernivtsi Medical Hospital, Chernivtsi
  - Dr. Olena Moroz, Dnipro
  - Dr. Pavlo Khaitov, Dnipro
  - Dr. Tamara Mishchenko, Kharkiv
  - Dr. Oleksandr Doroschenko, Krykhivtsi
  - Dr. Larysa Sokolova, Kyiv
  - Dr. Galusha, Kyiv
  - Dr. Olga Shulga, Lutsk
  - Dr.Tetyana Nehrych, Lviv
  - Dr. Svitlana Skhrobot, Ternopil
  - Dr. Sergii Moskovko, Vinnytsia